CLINICAL TRIAL: NCT01043224
Title: A Psoriasis Plaque Study Comparing Clobetasol Propionate Plus Calcipotriol Ointment With Clobetasol Propionate Ointment Alone, Calcipotriol Ointment Alone and a Vehicle Control for the Treatment of Psoriasis Vulgaris
Brief Title: A Psoriasis Plaque Test Comparing Products for the Treatment of Psoriasis Vulgaris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: PLQ-004; EudractCT No: 2009-012139-14 (Registry Identifier: European Clinical Trials Database)
Record Dates: First submitted 2010-01-05; First posted 2010-01-06 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2013-10

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Clobetasol propionate plus calcipotriol (Experimental)
  Interventions: Drug: Combination of clobetasol propionate plus calcipotriol ointment, clobetasol propionate ointment, calcipotriol ointment, and the ointment vehicle

INTERVENTIONS:
Drug: Combination of clobetasol propionate plus calcipotriol ointment, clobetasol propionate ointment, calcipotriol ointment, and the ointment vehicle — Once daily application

SUMMARY:
The purpose of this trial is to compare the anti-psoriatic effect of a topical combination product containing clobetasol propionate and calcipotriol in an ointment formulation to the single components in the same vehicle using a psoriasis plaque test design.

ELIGIBILITY:
Inclusion Criteria (in summary):

* Subjects having understood and signed an informed consent form
* Either sex
* Age 18 years or above
* All skin types and any ethnic origin
* Subjects with a diagnosis of psoriasis vulgaris with lesions located on arms, legs or trunk

Exclusion Criteria (in summary):

* Females who are pregnant, or who wish to become pregnant during the study, or who are breast feeding
* Systemic treatment with biological therapies (marketed or not marketed) with a possible effect on psoriasis vulgaris within 4 weeks (etanercept), 2 months (adalimumab, alefacept, infliximab), 4 months (ustekinmab) or 4 weeks/5 half-lives (which-ever is longer) for experimental biological products prior to randomisation
* Systemic treatments with all other therapies than biologicals, with a potential effect on psoriasis vulgaris (e.g., corticosteroids, vitamin D analogues, retinoids, immuno-suppressants) within the 4-week period prior to randomisation
* Subjects using one of the following topical drugs for the treatment of psoriasis within the 4 week period prior to randomisation

  * Potent or very potent (WHO group III-IV) corticosteroids
  * PUVA or Grenz ray therapy
* Subjects using one of the following topical drugs for the treatment of psoriasis within 2 weeks prior to randomisation

  * WHO group I-II corticosteroids
  * Topical retinoids
  * Vitamin D analogues
  * Topical immunomodulators (e.g. macrolides)
  * Anthracen derivatives
  * Tar
  * Salicylic acid
  * UVB therapy
* Subjects who have received treatment with any non-marketed drug substance (i.e., an agent which has not yet been made available for clinical use following registration) within the 4 week period prior to randomisation or longer, if the class of the substance requires a longer washout as defined above (e.g., biological treatments)
* Subjects with current participation in any other interventional clinical, based on interview of the subject
* Subjects with current diagnosis of guttate, erythrodermic, exfoliative or pustular psoriasis
* Subjects with known or suspected hypersensitivity to component(s) of the investigational products
* Subjects with known/suspected disorders of calcium metabolism associated with hypercalcaemia
* Subjects with known severe hepatic and/or severe renal insufficiency
* Subjects with any of the following conditions present on the plaque test areas: viral (e.g. herpes or varicella) lesions of the skin, fungal and bacterial skin infections, parasitic infections and atrophic skin
* Subjects with skin manifestations on the plaque test areas in relation to syphilis or tuberculosis, rosacea, perioral dermatitis, acne vulgaris, atrophic skin, striae atrophicae, fragility of skin veins, ichthyosis, acne rosacea, ulcers and wounds
* Subjects with any concomitant medical or dermatological disorder(s) which might preclude accurate evaluation of the psoriasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Total Clinical Score of clinical symptoms | 3 weeks

SECONDARY OUTCOMES:
Clinical scores, lesions thickness, NIR spectroscopic measurements | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Facy, PhD, Study Director — LEO Pharma
Locations (1):
- LEO Pharma investigational site, Nice, France

IPD SHARING:
Plan to Share IPD: No